CLINICAL TRIAL: NCT03003832
Title: A Cluster-randomized Trial of Modifying Electronic Health Record Defaults to Reduce the Prescribed Quantity of Opioid Analgesics in Primary Care and Emergency Department Settings
Brief Title: Electronic Defaults to Reduce Opioid Prescribing in Emergency Department and Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Marcus Bachhuber, Assistant Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-6036
Record Dates: First submitted 2016-12-06; First posted 2016-12-28 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention condition consists of a change to the electronic health record so that new opioid analgesic prescriptions automatically default to 10 pills (i.e., the "quantity dispensed" field is pre-populated). This value is modifiable by providers who can tailor the prescription based on clinical factors.
  Interventions: Other: Change in electronic health record default for new opioid analgesic prescriptions
- Standard of care (No Intervention): The control condition will be the usual electronic health record interface. The default number of pills varies by medication, most medications currently have either a blank default or a default of 30 pills.

INTERVENTIONS:
Other: Change in electronic health record default for new opioid analgesic prescriptions
  Arms: Intervention

SUMMARY:
The goal of this research is to investigate the impact of changing opioid analgesic prescribing defaults on the quantity of opioids prescribed for acute non-cancer pain in adult primary care and emergency department settings. We will change prescribing defaults for select short-acting opioid analgesics including immediate release oxycodone and hydrocodone as well as codeine and tramadol, including their co-formulations with acetaminophen. In a cluster-randomized trial of matched pairs of Montefiore Medical Center clinical sites, stratified by specialty and teaching status, we will evaluate the impact of this intervention on patient-level outcomes using 18 months of data (6 months pre-intervention and 12 months post-intervention).

ELIGIBILITY:
Clinical Site Inclusion Criteria:

* Primary care clinic (internal medicine, family medicine, or urgent care) or emergency department within Montefiore Medical Center

Patient Inclusion Criteria:

* Received a new opioid analgesic prescription, defined as no opioid analgesic prescription in the preceding 6 months

Patient Exclusion Criteria:

* Cancer diagnosis code within the past 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Initial prescription <= 10 pills (y/n) | Through study completion (18 months)
  Extracted from the electronic medical record

SECONDARY OUTCOMES:
Initial prescription number of pills | Through study completion (18 months)
  Extracted from the electronic medical record
Initial prescription morphine milligram equivalents | Through study completion (18 months)
  Extracted from the electronic medical record
Opioid analgesic re-order (y/n) | Within 30 days after the initial prescription
  Extracted from the electronic medical record
Total opioid analgesic pills prescribed, including re-orders | Within 30 days after the initial prescription
  Extracted from the electronic medical record
Total morphine milligram equivalents prescribed, including re-orders | Within 30 days after the initial prescription
  Extracted from the electronic medical record
Outpatient visits | Within 30 days after the initial prescription
  Extracted from the electronic medical record
Emergency department visits | Within 30 days after the initial prescription
  Extracted from the electronic medical record
Hospitalizations | Within 30 days after the initial prescription
  Extracted from the electronic medical record

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bachhuber MA, Nash D, Southern WN, Heo M, Berger M, Schepis M, Thakral M, Cunningham CO. Effect of Changing Electronic Health Record Opioid Analgesic Dispense Quantity Defaults on the Quantity Prescribed: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e217481. doi: 10.1001/jamanetworkopen.2021.7481. PMID 33885773
- [Derived] Bachhuber MA, Nash D, Southern WN, Heo M, Berger M, Schepis M, Cunningham CO. Reducing the default dispense quantity for new opioid analgesic prescriptions: study protocol for a cluster randomised controlled trial. BMJ Open. 2018 Apr 20;8(4):e019559. doi: 10.1136/bmjopen-2017-019559. PMID 29678969